CLINICAL TRIAL: NCT05549843
Title: Safety and Efficacy of Manual Therapy in the Treatment of Hemophilic Arthropathy of the Ankle. A Pilot Study
Brief Title: Manual Therapy in the Treatment of Hemophilic Arthropathy of the Ankle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: He-AnklePilot
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemophilia group (Experimental): Intervention protocol:
  * Preparatory work: active mobilizations with the patient supine.
  * Global passive mobilization of the forefoot and midfoot.
  * Calcaneocuboid mobilization, functional and structural work of said joint.
  * Astragaloscaphoid mobilization, functional and structural work of said joint.
  * Talar manipulation dorsally.
  * Manipulation-tibial displacement:
  * Tibiotarsal decompression: 2 very gentle high-speed and short-course tibial-tarsal manipulations.
  * Plantar fascia induction for foot captors of the plantar fascia.
  * Tibiotarsal sustained traction technique (unwinding)
  * Sural triceps induction technique:
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — Each session will last approximately 50-60 minutes, with 1 physiotherapy session per week over a period of 3 weeks. Each session is made up of 10 steps, of which 9 correspond to manual interventions commonly used in the field of manual therapy.

SUMMARY:
Introduction: Hemophilic ankle arthropathy is manifested by degenerative functional alterations (deficit of muscle strength, mobility and proprioception), intra-articular alterations and chronic pain. Manual therapy techniques are used to treat soft tissue adhesions, relieve pain and reduce tissue sensitivity.

Design. randomized pilot trial. Aimed: To evaluate the safety and effectiveness of a protocol by manual therapy techniques in patients with hemophilic ankle arthropathy.

Patients: 24 patients with ankle arthropathy will be recruited for inclusion in the study. Patients will be recruited in seven centers, from different regions of Spain.

Intervention: Each session will last approximately 50-60 minutes, with 1 physiotherapy session per week for a period of 3 weeks. Patients will be evaluated at baseline, after the intervention, and after a follow-up period of 3 weeks. The treatment program includes 10 exercises that must be administered bilaterally.

Measuring instruments and study variables: Visual Analog Scale and pressure algometer (joint pain); Leg motion (ankle range of motion); and Haemophilia Joint Health Score (joint health). At the same time, the study will allow to determine joint bleeding caused by applied physiotherapy treatment.

Expected results: To demonstrate the safety of this Physiotherapy technique in patients with hemophilia. Likewise, an improvement in ankle pain, joint motion, joint health and pressure pain threshold.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* With severe (<1% FVIII/FIX) or moderate (1-5% FVIII/FIX) phenotype of hemophilia
* Over 18 years
* With medical diagnosis of ankle arthropathy and with clinical evaluation by Hemophilia Joint Health Score
* In prophylactic treatment with FVIII / FIX concentrates for coagulation

Exclusion Criteria:

* Patients with inhibitors (antibodies against FVIII or FIX)
* Patients with neurological or cognitive disorders that prevent the understanding of questionnaires and physical tests
* Failure to sign the informed consent document

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-02-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline frequency of ankle hemarthrosis after treatment and at 3 weeks | Screening visit, within the first seven days after treatment and after two months follow-up
  Weekly follow-up by telephone calls in the experimental phase. The evaluator will conduct a survey with closed questions and answers on the clinical manifestations of hemarthrosis to rule out joint or muscle bleeding. The frequency of hemarthrosis will be measured with the total number of bleedings in the study period in each evaluation.

SECONDARY OUTCOMES:
Change from baseline ankle joint pain after treatment and at 3 weeks | Screening visit, within the first seven days after treatment and after two months follow-up
  Visual analogic scale (VAS). This scale will be used to evaluate the perception of joint pain, where ankle joint pain ranges from 0 to 10 points (no pain to maximum perceived pain).
Change from baseline pressure pain threshold of ankle after treatment and at 3 weeks | Screening visit, within the first seven days after treatment and after two months follow-up
  Pressure algometer. Measuring instrument used to evaluate pressure joint pain. The instrument shall consist of a measuring device attached to a hard rubber tip 1.1 cm in diameter. Its sphere shall be calibrated in kg/cm2 with divisions of 0.1 kg/cm2. The pressure algometry methodology applied was based mainly on the study by Hogeweg.
  Before taking the measurements, patients will be instructed to say "yes" as soon as pressure exerted by the algometer becomes slightly unpleasant. The pressure algometer shall be kept perpendicular to the surface of the skin with the right hand, stabilizing the axis of the instrument using the thumb and index finger of the left hand. The pressure shall be increased at a uniform rate of approximately 1 kg/cm2 per second. As soon as the subject, according to the instructions, says "yes", the pressure will be stopped and the score will be noted.
Change from baseline ankle joint damage after treatment and at 3 weeks | Screening visit, within the first seven days after treatment and after two months follow-up
  Hemophilia Joint Health Score (HJHS). This measuring instrument will be used to evaluate the joint condition of ankles. It includes 8 items (inflammation and its duration, pain, atrophy and muscle strength, crepitus, and reduced flexion and extension) ranging from 0 to 20 points per joint (the higher the score, the greater the joint deterioration).
Change from baseline ankle range of motion after treatment and at 3 weeks | Screening visit, within the first seven days after treatment and after two months follow-up
  Leg motion device. The test will be conducted in accordance with the procedures for conducting the weight-bearing lunge test. The subjects will stand to assess, in the Leg Motion system, with the big toe on the starting line and the knee touching a metal stick. While patients hold the position, they will be instructed on how to perform a lunge in which the knee will be flexed with the aim of touching a metal rod with its anterior part. The metal rod will move away from the foot up to the maximum ankle dorsiflexion allowed, without taking the heel off the ground and with knee contact on the rod. Maximum dorsiflexion ROM will be defined as the maximum distance from the toe to the metal rod while maintaining contact with the knee for three seconds, without lifting the heel. Three measurements will be made for each ankle and the mean value will be used for data analysis. All measurements will be made with the patient barefoot, first with one leg and then with the contralateral leg.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Truque-Diaz C, Merono-Gallut J, Cuesta-Barriuso R, Perez-Llanes R. Joint and Myofascial Manual Therapy Techniques in Haemophilic Ankle Arthropathy: A Randomized Pilot Study. Haemophilia. 2025 Mar;31(2):295-303. doi: 10.1111/hae.70002. Epub 2025 Feb 7. PMID 39917949